CLINICAL TRIAL: NCT00120185
Title: Study of the Immunological Efficacy of Using Subcutaneous Interleukin-2 (IL-2) in Antiretroviral Naïve HIV-1-Infected Subjects With a CD4 Cell Count Above 300/mm3. ANRS 119 Trial INTERSTART
Brief Title: Efficacy of Using Interleukin-2 in Antiretroviral Naïve HIV Patients (ANRS119)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Chiron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-003897-27; ANRS119 Interstart
Record Dates: First submitted 2005-07-08; First posted 2005-07-15 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: HIV Infections
Keywords: HIV Infections; Interleukin-2
MeSH Terms: conditions — HIV Infections | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Interleukin-2

SUMMARY:
Interleukin-2 (IL-2) increases the number of CD4 cells in HIV-1 infected patients under highly active antiretroviral therapy (HAART) with a CD4 cell count over 200/mm3, but its activity in patients without antiretroviral therapy is unknown. This study will test the efficacy and safety of IL-2 in naïve patients with a CD4 count between 300 and 500/m3.

DETAILED DESCRIPTION:
IL-2 is produced naturally in the body and helps CD4 cells multiply. In earlier studies in HIV-infection, most of the patients with a controlled viral load under antiretroviral therapy and a high level of CD4 cell count (over 200/mm3) who received IL-2, experienced an increase of their CD4 cell count superior to what is observed with antiretroviral therapy alone. The efficacy of IL-2 when the viral load is high and the patient is not receiving antiretroviral therapy is not known. The purpose of this multicentric national study is to compare the effects of IL-2 versus no treatment in HIV naïve patients. One hundred thirty HIV-1-infected patients, with a CD4 count between 300 and 500/mm3, will be randomly assigned to one of two treatment groups : IL-2 or no treatment. The group with IL-2 will receive a dose of 4.5 million international units by subcutaneous injection twice a day for 5 days (up to a total of 5 cycles, ending at Week 96), the first three cycles 8 weeks apart. Evaluation will be done at week 96. The primary endpoint is the proportion of patients reaching an absolute CD4 count below 300/mm3 at Week 96. Secondary endpoints include the occurrence of HIV-related events, drug safety and the evolution of CD4 cells and of HIV RNA and HIV DNA loads over time.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with proven HIV-1-infection
* No prior exposition to antiretrovirals
* CD4 cell count between 300 and 500/mm3
* Signed written inform consent

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2003-12; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reaching an absolute CD4 count below 300/mm3 at W96

SECONDARY OUTCOMES:
Group B or C events (1993 CDC classification of HIV infection)
Initiation of antiretroviral therapy
Evolution of the CD4 count during the study
Time to the first visit with a CD4 count below 300/mm3
Tolerance of IL-2
Evolution of the plasma HIV RNA load
Evolution of the HIV DNA level in PBMCs
Quality of life at W96
Assessment of lipodystrophy at W96
Immunological substudies (CD4 homeostasis, anti HIV cellular immune responses) at W96

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Molina, MD, Principal Investigator — Hopital Saint Louis Paris service des Maladies infectieuses et Tropicales; Jean-Pierre Aboulker, MD, Study Chair — Inserm SC10
Locations (1):
- Service des Maladies Infectieuses, Paris, France

REFERENCES:
- [Derived] Molina JM, Levy Y, Fournier I, Hamonic S, Bentata M, Beck-Wirth G, Gougeon ML, Venet A, Madelaine I, Sereni D, Jeanblanc F, Boulet T, Simon F, Aboulker JP; Agence Nationale de Recherches sur le SIDA et les Hepatites Virales (ANRS) 119 Interstart Study Team. Interleukin-2 before antiretroviral therapy in patients with HIV infection: a randomized trial (ANRS 119). J Infect Dis. 2009 Jul 15;200(2):206-15. doi: 10.1086/599989. PMID 19508157